CLINICAL TRIAL: NCT06146998
Title: Development of 3D Printing High-Fidelity Thyroid Fine Needle Aspiration Exam Medical Education Model to Facilitate Patient Education
Brief Title: Three-dimensional Thyroid Education Model
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fu Jen Catholic University (Other)
Responsible Party: Principal Investigator, Ke-Yun, Chao, Group leader of Respiratory Therapists, Fu Jen Catholic University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: FJUH111215
Record Dates: First submitted 2023-11-20; First posted 2023-11-27 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Satisfaction, Patient
Keywords: 3D printing; medical education model; high-fidelity simulation; thyroid; fine needle aspiration
MeSH Terms: conditions — Patient Satisfaction; Thyroid Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D model group (Experimental): Received a explanation combined with 3D medical education model
  Interventions: Other: 3D health education model
- traditional explanation group (Active Comparator): Received a regular explanation
  Interventions: Other: Verbal explanation

INTERVENTIONS:
Other: 3D health education model — explanation combined with 3D health education model
  Arms: 3D model group
Other: Verbal explanation — Regular explanation
  Arms: traditional explanation group

SUMMARY:
The purpose of our study is to develop a high-fidelity thyroid education model, that can be utilized for patient education. This model can assist them in gaining a better understanding of the thyroid's structure, providing patients with insights into their own conditions and thyroid fine needle aspiration examinations.

DETAILED DESCRIPTION:
Background： Thyroid nodular disorder is one of the most common diseases in Endocrine clinics. And thyroid fine needle aspiration examination is the most important exam in evaluating the nature of thyroid nodules. In previous studies, 3D thyroid models have been introduced for patient education before thyroid surgery. Nevertheless, thyroid models that can be used to practice thyroid fine needle aspiration examination were scarce.

Study Design： This is a prospective study.

Methods： In our study, 3D printing technology will be used to create the thyroid high-fidelity model. We plan to choose 3D printing materials that explain thyroid fine needle aspiration for patient education efficacy evaluation.

Effect： Through the creation of this thyroid fine needle aspiration model, we hope to enhance patients' comprehension of the thyroid and thyroid nodules. The results of our study could be applied in hospitals to improve patient education.

Key words： 3D printing; medical education model; high-fidelity simulation; thyroid; fine needle aspiration

ELIGIBILITY:
Inclusion Criteria:

* Thyroid nodule detected
* Thyroid ultrasound-guided fine-needle aspiration is needed

Exclusion Criteria:

* Previously underwent thyroid ultrasound-guided fine-needle aspiration
* Refused to participate in the study

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Medical education effectiveness questionnaire | immediately after the intervention
  higher means a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Ke-Yun Chao, PhD, Principal Investigator — Fu Jen Catholic University Hospital
Locations (1):
- Fu Jen Catholic University Hospital, Fu Jen Catholic University, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No